CLINICAL TRIAL: NCT03712449
Title: Canada Global HARMONY: Prospective, Multi-site, Study to Evaluate Subject Satisfaction With Facial Appearance Overall and the Aesthetic and Psychosocial Impact of Combined Facial Treatment
Brief Title: A Study to Evaluate Participant Satisfaction With Facial Appearance Overall and the Aesthetic and Psychosocial Impact of Combined Facial Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMO-MA-FAS-0579
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Results first posted 2021-08-25 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Facial Rhytides, Skin Folds, Loss of Volume and Skin Quality
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- BELKYRA Treatment (Experimental): BELKYRA was injected into the subcutaneous fat for maximum of 6 treatments, 1 month apart from Month 0 to Month 5. Maximum dose did not exceed 100 milligrams (mg) [10 milliliters (mL)] in a single treatment.
  SkinMedica products: (Facial Cleanser, TNS Essential Serum®, Rejuvenative Moisturizer, Optional: Total Defense + Repair Broad Spectrum Sunscreen SPF34), applied daily from Month 6 to Month 11.
  Facial filler injectable treatment (JUVÉDERM VOLBELLA with Lidocaine and/or JUVÉDERM VOLIFT with Lidocaine and/or JUVÉDERM VOLUMA with Lidocaine and/or JUVÉDERM VOLITE with Lidocaine) from Month 6 to Month 8. The volume of filler injected at initial and touch-up treatments was determined by the investigator.
  BOTOX Cosmetic 20 units (U) to glabellar lines and/or 2-6 U injected bilaterally to crow's feet lines and/or 24 U total injected to forehead lines at Month 9 and Month 10.
  Interventions: Device: JUVÉDERM®; Drug: BOTOX Cosmetic®; Drug: BELKYRA®; Other: SkinMedica
- Non-BELKYRA Treatment (Experimental): Participants who did not receive BELKYRA.
  SkinMedica products: (Facial Cleanser, TNS Essential Serum®, Rejuvenative Moisturizer, Optional: Total Defense + Repair Broad Spectrum Sunscreen SPF34), applied daily from Month 0 to Month 5.
  Facial filler injectable treatment (JUVÉDERM VOLBELLA with Lidocaine and/or JUVÉDERM VOLIFT with Lidocaine and/or JUVÉDERM VOLUMA with Lidocaine and/or JUVÉDERM VOLITE with Lidocaine) from Month 0 to Month 2. The volume of filler injected at initial and touch-up treatments was determined by the investigator.
  BOTOX Cosmetic 20 units (U) to glabellar lines and/or 2-6 U injected bilaterally to crow's feet lines and/or 24 U total injected to forehead lines at Month 3 and Month 4.
  Interventions: Device: JUVÉDERM®; Drug: BOTOX Cosmetic®; Other: SkinMedica

INTERVENTIONS:
Device: JUVÉDERM® — Facial filler injection (JUVÉDERM VOLBELLA with Lidocaine, and/or JUVÉDERM VOLIFT with Lidocaine, and/or JUVÉDERM VOLUMA with Lidocaine, and/or JUVÉDERM VOLITE with Lidocaine) from Month 6 to Month 8 (BELKYRA Treatment) and Month 0 to Month 2 (Non-BELKYRA Treatment).
Drug: BOTOX Cosmetic® — BOTOX Cosmetic, 20 U to glabellar lines and/or 2-6 U injected bilaterally to crow's feet lines and/or 24 U injected to forehead lines at Month 9 and Month 10 (BELKYRA Treatment) and at Month 3 and Month 4 (Non-BELKYRA Treatment).
Drug: BELKYRA® — BELKYRA, subcutaneous injection for maximum of 6 treatments, 1 month apart from Month 0 to Month 5. Maximum dose = 100 mg (10mL).
  Arms: BELKYRA Treatment
Other: SkinMedica — SkinMedica products (Facial Cleanser, TNS Essential Serum®, Rejuvenative Moisturizer, Optional: Total Defense + Repair Broad Spectrum Sunscreen SPF34), applied daily from Month 6 to Month 11 (BELKYRA Treatment) and Month 0 to Month 5 (Non-BELKYRA Treatment).

SUMMARY:
The objective of this study is to quantify the psychological and emotional impact of comprehensive aesthetic treatment with a portfolio of Allergan products by measuring the change in participant's satisfaction with facial appearance from baseline to the final study visit.

ELIGIBILITY:
Inclusion Criteria:

* Accept the obligation not to receive any other facial procedures or treatments at any time during the study that are not related to the study
* Women of childbearing potential must have a negative urine pregnancy test before each injectable treatment and practice a reliable method of contraception throughout the study
* Willing to avoid direct and prolonged sun exposure to the facial skin, which includes tanning beds, for the duration of the study

Exclusion Criteria:

* History of any intervention to treat submental fat (SMF) (e.g. liposuction, surgery, or lipolytic agents)
* History of trauma associated with the chin or neck areas that in the judgment of the investigator may affect evaluation of safety or efficacy of treatment
* An anatomical feature (e.g. predominant subplatysmal fat, loose skin in the neck or chin area, prominent platysmal bands) for which reduction in SMF may, in the judgment of the investigator, result in an aesthetically unacceptable outcome
* Evidence of any cause of enlargement in the submental area (e.g. thyroid enlargement, cervical adenopathy, ptotic submandibular gland) other than localized SMF
* Any medical condition (e.g. respiratory, cardiovascular, hepatic, neurological disease, or thyroid dysfunction) that would interfere with assessment of safety or efficacy or compromise the participant's ability to undergo study procedures or give informed consent
* Body mass index (BMI) > 30
* Known allergy or sensitivity to the study products or their components
* Pregnant, lactating, or planning to become pregnant at any time during the study
* Received BOTOX Cosmetic® or treatment with any other botulinum toxin product for any condition at any time prior to entry in the study
* Received (or is planning to receive) anticoagulation, antiplatelet or thrombolytic medications (e.g. warfarin) or other substances known to increase coagulation time from 10 days prior to injection and up to 3 days post-injection
* Undergone plastic surgery of the face and/or neck, tissue grafting, or tissue augmentation with silicone, fat, or other permanent dermal fillers, or be planning to undergo any of these procedures at any time during the study
* Received temporary or semi-permanent facial or neck dermal filler injections (e.g. hyaluronic acid (HA), calcium hydroxylapatite, L-polylactic acid) at any time prior to entry in the study
* Received mesotherapy, skin resurfacing (laser, photomodulation, intense pulsed light, radio frequency, dermabrasion, chemical peel, or non-ablative procedures) in the face or neck within 6 months prior to study enrollment
* Began use of any new over-the-counter (OTC) or prescription, oral or topical, antiwrinkle products on the facial area within 90 days prior to enrollment or planning to begin use of such products at any time during the study
* Lip tattoos, facial hair or scars that would interfere with visualization of the lips and perioral area for the effectiveness assessments
* Received any investigational product within 60 days prior to study enrollment or planning to participate in another investigation during the course of this study
* An employee (or a relative of an employee) of the investigators, Allergan, or representative of Allergan
* Current use of oral corticosteroids
* Current use of nonsteroidal anti-inflammatory drugs (NSAIDs) (e.g. aspirin, ibuprofen) with the exception of a daily low dose of aspirin, from 10 days prior to injection up to 3 days post-injection
* Prescription topical retinoid therapy and/or topical hormone cream applied to the face, for potential participants who have not been on a consistent dose regimen for at least 6 months prior to enrollment and who are unable to maintain regimen for the study
* Systemic retinoid therapy within one year prior to study enrollment
* Medical condition that may increase the risk of exposure to botulinum toxin including diagnosed myasthenia gravis, Eaton-Lambert Syndrome, amyotrophic lateral sclerosis, or any other disease that might interfere with neuromuscular function
* Current use of aminoglycoside antibiotics, curare-like agents, or agents that might interfere with neuromuscular (skeletal) function
* History of facial nerve palsy
* Anticipated need for treatment with botulinum toxin of any serotype for any reason during the study (other than study treatment)
* Tendency to accumulate fluid in the lower eyelids, or large infraorbital fat pads, i.e., significant convexity or projection from the infraorbital fat pads
* Mid-face volume deficit due to congenital defect, trauma, abnormalities in adipose tissue related to immune-mediated diseases such as generalized lipodystrophy (e.g. juvenile dermatomyositis), partial lipodystrophy (e.g. Barraquer-Simons syndrome), inherited disease, or human immunodeficiency virus-related disease
* Undergone oral surgery or other dental procedures (e.g. tooth extraction, orthodontia, or implantation) within 30 days prior to enrollment or be planning to undergo any of these procedures during the study
* Participants with neuromuscular disorders including generalized muscle weakness, diplopia, ptosis, dysphonia, dysarthria, severe dysphagia, and respiratory compromise
* Participants with a history of allergies or hypersensitivity to HA or lidocaine

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Sangha, Study Director — Allergan
Locations (7):
- Canada (7):
  - Carruthers & Humphrey Cosmetic Dermatology, Vancouver, British Columbia
  - Shannon Humphrey, Vancouver, British Columbia
  - Project Skin MD Vancouver, Vancouver, British Columbia
  - Pacific Derm, Vancouver, British Columbia
  - Dermetics, Burlington, Ontario
  - Dr Nowell Solish, Toronto, Ontario
  - Bertucci MedSpa, Woodbridge, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 59 participants were enrolled, of which 58 were randomized in the study to receive BELKYRA and non-BELKYRA treatment in the ratio of approximately 1:2. Participants receiving BELKYRA treatment entered the study at Month 0 continuing on to Month 11. Participants not receiving BELKYRA following screening entered the study at Month 0 (similar to Month 6 visit of the BELKYRA arm) to begin treatment with JUVÉDERM hyaluronic acid (HA) facial fillers, SkinMedica, and BOTOX Cosmetic.
Groups:
- BELKYRA Treatment: BELKYRA was injected into the subcutaneous fat for maximum of 6 treatments, 1 month apart from Month 0 to Month 5. Maximum dose did not exceed 100 mg [10 mL] in a single treatment.
  SkinMedica products: (Facial Cleanser, TNS Essential Serum®, Rejuvenative Moisturizer, Optional: Total Defense + Repair Broad Spectrum Sunscreen SPF34), applied daily from Month 6 to Month 11.
  Facial filler injectable treatment (JUVÉDERM VOLBELLA with Lidocaine and/or JUVÉDERM VOLIFT with Lidocaine and/or JUVÉDERM VOLUMA with Lidocaine and/or JUVÉDERM VOLITE with Lidocaine) from Month 6 to Month 8. The volume of filler injected at initial and touch-up treatments was determined by the investigator.
  BOTOX Cosmetic 20 units (U) to glabellar lines and/or 2-6 U injected bilaterally to crow's feet lines and/or 24 U total injected to forehead lines at Month 9 and Month 10.
Period: Overall Study
Arm/Group | BELKYRA Treatment | Non-BELKYRA Treatment
Started | 13 | 46
Full Analysis Population (Full Analysis Population included all participants who had met all eligibility criteria at the screening visit and received any product used as treatment in this study.) | 13 | 45
Completed | 13 | 45
Not Completed | 0 | 1
Not completed — Withdraw Consent | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Population included all participants who had met all eligibility criteria at the screening visit and received any product used as treatment in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | BELKYRA Treatment | Non-BELKYRA Treatment | Total
Number analyzed (Participants) | 13 | 45 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (3.88) | 51.4 (7.93) | 51.8 (7.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 40 | 51
  Male | 2 | 5 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Rasch-transformed Score of FACE-Q Satisfaction With Facial Appearance Overall Scale to End of Study
Description: The participant assessed satisfaction using the 10 items on the FACE-Q: Satisfaction with Facial Appearance questionnaire measured on a 4-point scale where 1=very dissatisfied, 2=somewhat dissatisfied, 3=somewhat satisfied, and 4=very satisfied. The responses to the items were converted to a 100-point Rasch transformed scale score with 0 (worst) to 100 (best). Higher scores indicate higher satisfaction. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Prior to Treatment) to End of Study (BELKYRA Treatment: Up to Month 11; Non-BELKYRA Treatment: Up to Month 5)
Population: Evaluable Population included all participants as defined in the Full Analysis Population who had at least one post treatment efficacy assessment at the final visit. Full Analysis Population included all participants who had met all eligibility criteria at the screening visit and received any product used as treatment in this study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BELKYRA Treatment | Non-BELKYRA Treatment
Number analyzed (Participants) | 13 | 45
score on a scale
  Baseline | 40.9 (16.79) | 37.8 (10.96)
  Change from Baseline to End of Study | 21.5 (17.76) | 32.9 (17.40)
Statistical Analysis 1: Comparison: BELKYRA Treatment; Test type: Other — The data was analyzed using Paired t-test. If normality was not met, then the Wilcoxon signed-rank test was used; p = 0.0009, Paired t-test/Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: Non-BELKYRA Treatment; Test type: Other — The data was analyzed using Paired t-test. If normality was not met, then the Wilcoxon signed-rank test was used; p < 0.0001, Paired t-test/Wilcoxon Signed Rank Test

2. Secondary Outcome: Change From Baseline in Participant's Assessment of Expectations of Life Change as Measured by Rasch-transformed Score of FACE-Q Expectations Scale to End of Study
Description: The participant assessed expectations of life change using the FACE-Q questionnaire measured on a 4-point expectations scale where 1=definitely disagree, 2=somewhat disagree, 3=somewhat agree, 4=definitely agree. The responses to the items on the questionnaire were converted to a 100-point Rasch transformed scale score with 0 (worst) to 100 (best). A positive change from Baseline indicates improvement.
Time Frame: Baseline (Prior to Treatment) to End of Study (BELKYRA Treatment: Up to Month 11; Non-BELKYRA Treatment: Up to Month 5)
Population: Evaluable Population included all participants as defined in the Full Analysis Population who had at least one post treatment efficacy assessment at the final visit. Full Analysis Population included all participants who had met all eligibility criteria at the screening visit and received any product used as treatment in this study. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BELKYRA Treatment | Non-BELKYRA Treatment
Number analyzed (Participants) | 13 | 45
score on a scale
  Baseline | 51.0 (12.96) | 50.1 (12.24)
  Change from Baseline to End of Study: number analyzed (Participants) | 6 | 28
  Change from Baseline to End of Study | -1.3 (11.50) | 4.8 (11.48)
Statistical Analysis 1: Comparison: BELKYRA Treatment; Test type: Other — The data was analyzed using Paired t-test. If normality was not met, then the Wilcoxon signed-rank test was used; p = 0.7878, Paired t-test/Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: Non-BELKYRA Treatment; Test type: Other — The data was analyzed using Paired t-test. If normality was not met, then the Wilcoxon signed-rank test was used; p = 0.0349, Paired t-test/Wilcoxon Signed Rank Test

3. Secondary Outcome: Change From Baseline in Participant's Assessment of Age-related Facial Appearance as Measured by Rasch-transformed Score of FACE-Q Aging Appraisal Scale to End of Study
Description: The participant assessed age-related facial appearance using the FACE-Q questionnaire measured on a 4-point aging appraisal scale where 1=definitely disagree, 2=somewhat disagree, 3=somewhat agree, 4=definitely agree. The responses to the items on the questionnaire were converted to a 100-point Rasch transformed scale score. Lower scores indicated better outcome and responders were defined as having achieved a younger category. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Prior to Treatment) to End of Study (BELKYRA Treatment: Up to Month 11; Non-BELKYRA Treatment: Up to Month 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BELKYRA Treatment | Non-BELKYRA Treatment
Number analyzed (Participants) | 13 | 45
score on a scale
  Baseline | 41.7 (17.66) | 40.4 (21.73)
  Change from Baseline to End of Study | 23.1 (23.72) | 35.6 (21.43)
Statistical Analysis 1: Comparison: BELKYRA Treatment; Test type: Other — The data was analyzed using Paired t-test. If normality was not met, then the Wilcoxon signed-rank test was used; p = 0.0043, Paired t-test/Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: Non-BELKYRA Treatment; Test type: Other — The data was analyzed using Paired t-test. If normality was not met, then the Wilcoxon signed-rank test was used; p < 0.0001, Paired t-test/Wilcoxon Signed Rank Test

4. Secondary Outcome: Change From Baseline in Participant's Assessment of Psychological Well-being as Measured by Rasch-transformed Score of FACE-Q Psychological Function Scale to End of Study
Description: The participant assessed psychological well-being using the FACE-Q questionnaire measured on a 4-point psychological function scale where 1=definitely disagree, 2=somewhat disagree, 3=somewhat agree, 4=definitely agree. The responses to the items on the questionnaire were converted to a 100-point Rasch transformed scale score with 0 (worst) to 100 (best). Higher scores indicate higher well-being. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Prior to Treatment) to End of Study (BELKYRA Treatment: Up to Month 11; Non-BELKYRA Treatment: Up to Month 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BELKYRA Treatment | Non-BELKYRA Treatment
Number analyzed (Participants) | 13 | 45
score on a scale
  Baseline | 57.6 (24.09) | 67.6 (23.79)
  Change from Baseline to End of Study | 21.3 (19.16) | 18.0 (22.02)
Statistical Analysis 1: Comparison: BELKYRA Treatment; Test type: Other — The data was analyzed using Paired t-test. If normality was not met, then the Wilcoxon signed-rank test was used; p = 0.0017, Paired t-test/Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: Non-BELKYRA Treatment; Test type: Other — The data was analyzed using Paired t-test. If normality was not met, then the Wilcoxon signed-rank test was used; p < 0.0001, Paired t-test/Wilcoxon Signed Rank Test

5. Secondary Outcome: Change From Baseline in Participant's Assessment of Social Function as Measured by Rasch-transformed Score of FACE-Q Social Function Scale to End of Study
Description: The participant assessed social function using the FACE-Q questionnaire measured on a 4-point social function scale where 1=definitely disagree, 2=somewhat disagree, 3=somewhat agree, 4=definitely agree. The responses to the items on the questionnaire were converted to a 100-point Rasch transformed scale score with 0 (worst) to 100 (best). Higher scores indicate higher social function. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Prior to Treatment) to End of Study (BELKYRA Treatment: Up to Month 11; Non-BELKYRA Treatment: Up to Month 5)
Population: Evaluable Population included all participants as defined in the Full Analysis Population who had at least one post treatment efficacy assessment at the final visit. Full Analysis Population included all participants who had met all eligibility criteria at the screening visit received any product used as treatment in this study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BELKYRA Treatment | Non-BELKYRA Treatment
Number analyzed (Participants) | 13 | 45
score on a scale
  Baseline | 54.8 (20.84) | 63.1 (18.46)
  Change from Baseline to End of Study | 18.6 (22.17) | 15.4 (20.74)
Statistical Analysis 1: Comparison: BELKYRA Treatment; Test type: Other — The data was analyzed using Paired t-test. If normality was not met, then the Wilcoxon signed-rank test was used; p = 0.0105, Paired t-test/Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: Non-BELKYRA Treatment; Test type: Other — The data was analyzed using Paired t-test. If normality was not met, then the Wilcoxon signed-rank test was used; p < 0.0001, Paired t-test/Wilcoxon Signed Rank Test

6. Secondary Outcome: Change From Baseline in Participant's Assessment of Overall Satisfaction With Skin as Measured by Rasch-transformed Score of FACE-Q Satisfaction With Skin Scale to End of Study
Description: The participant assessed overall satisfaction with skin using the FACE-Q questionnaire measured on a 4-point scale where 1=very dissatisfied, 2=somewhat dissatisfied, 3=somewhat satisfied, and 4=very satisfied. The responses to the items on the questionnaire were converted to a 100-point Rasch transformed scale score with 0 (worst) to 100 (best). Higher scores indicate higher satisfaction. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Prior to Treatment) to End of Study (BELKYRA Treatment: Up to Month 11; Non-BELKYRA Treatment: Up to Month 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BELKYRA Treatment | Non-BELKYRA Treatment
Number analyzed (Participants) | 13 | 45
score on a scale
  Baseline | 38.5 (17.61) | 36.3 (17.14)
  Change from Baseline to End of Study | 21.6 (19.62) | 34.2 (18.53)
Statistical Analysis 1: Comparison: BELKYRA Treatment; Test type: Other — The data was analyzed using Paired t-test. If normality was not met, then the Wilcoxon signed-rank test was used; p = 0.0004, Paired t-test/Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: Non-BELKYRA Treatment; Test type: Other — The data was analyzed using Paired t-test. If normality was not met, then the Wilcoxon signed-rank test was used; p < .0001, Paired t-test/Wilcoxon Signed Rank Test

7. Secondary Outcome: Number of Participants With Participant's Assessment of Age-related Facial Appearance as Measured by Self-perception of Age (SPA) Questionnaire (Item 1)
Description: The participant assessed age-related facial appearance using the 3 items on the SPA Questionnaire. Participants were asked 'how they think of their facial appearance looks compared to their age on the day of assessment' and participants had to respond in any one of the following responses: 1) I look my current age, or 2) I look (enter number of years) years younger, or 3) I look (enter number of years) years older. Item 1: Number of participants who responded 'I look my current age' is reported.
Time Frame: Baseline (Prior to Treatment) to End of Study (BELKYRA Treatment: Up to Month 11; Non-BELKYRA Treatment: Up to Month 5)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BELKYRA Treatment | Non-BELKYRA Treatment
Number analyzed (Participants) | 13 | 45
Participants
  Look Current Age; Baseline | 3 | 25
  Look Current Age; End of Study | 2 | 10

8. Secondary Outcome: Change From Baseline in Participant's Assessment of Age-related Facial Appearance as Measured by SPA Questionnaire (Items 2 and 3) to End of Study
Description: The participant assessed age-related facial appearance using the 3 items on the SPA Questionnaire. Participants were asked 'how they think of their facial appearance looks compared to their age on the day of assessment' and participants had to respond in any one of the following responses: 1) I look my current age, or 2) I look (enter number of years) years younger, or 3) I look (enter number of years) years older. Results for Items 2 and 3 are reported. The higher number of years in Item 2 implies better self-perception of age; a positive change from Baseline indicates improvement. The fewer number of years in Item 3 implies better self-perception of age; a negative change from Baseline indicates improvement.
Time Frame: Baseline (Prior to Treatment) to End of Study (BELKYRA Treatment: Up to Month 11; Non-BELKYRA Treatment: Up to Month 5)
Population: as for outcome 2
Measure: Median (Full Range); unit: years
Arm/Group | BELKYRA Treatment | Non-BELKYRA Treatment
Number analyzed (Participants) | 13 | 45
years
  Look (Number of Years) Younger; Baseline: number analyzed (Participants) | 3 | 10
  Look (Number of Years) Younger; Baseline | 3.0 [2 to 5] | 5.0 [3 to 10]
  Look (Number of Years) Younger; Change from Baseline to End of Study: number analyzed (Participants) | 3 | 10
  Look (Number of Years) Younger; Change from Baseline to End of Study | 6.0 [-1 to 10] | 2.5 [0 to 8]
  Look (Number of Years) Older; Baseline: number analyzed (Participants) | 7 | 10
  Look (Number of Years) Older; Baseline | 5.0 [2 to 10] | 5.5 [5 to 10]
  Look (Number of Years) Older; Change from Baseline to End of Study: number analyzed (Participants) | 2 | 1
  Look (Number of Years) Older; Change from Baseline to End of Study | -2.5 [-5 to 0] | -5.0 [-5 to -5]

9. Secondary Outcome: Number of Participants by Global Aesthetic Improvement Scale (GAIS) Categories as Assessed by the Investigator
Description: The investigator assessed the participant's improvement from Baseline to the End of Study using the GAIS where: 2=Much Improved, 1=Improved, 0=No Change, -1=Worse and -2=Much Worse.
Time Frame: Baseline (Prior to Treatment) to the End of Study (BELKYRA Treatment: Up to Month 11; Non-BELKYRA Treatment: Up to Month 5)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BELKYRA Treatment | Non-BELKYRA Treatment
Number analyzed (Participants) | 13 | 45
Participants
  2=Much Improved | 11 | 42
  1=Improved | 2 | 3
  0=No Change | 0 | 0
  -1=Worse | 0 | 0
  -2=Much Worse | 0 | 0

10. Secondary Outcome: Number of Participants by Global Aesthetic Improvement Scale (GAIS) Categories as Assessed by the Participant
Description: The participants self-assessed their improvement from Baseline to the End of Study using the GAIS where: 2=Much Improved, 1=Improved, 0=No Change, -1=Worse and -2=Much Worse.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BELKYRA Treatment | Non-BELKYRA Treatment
Number analyzed (Participants) | 13 | 45
Participants
  2=Much Improved | 11 | 33
  1=Improved | 2 | 11
  0=No Change | 0 | 1
  -1=Worse | 0 | 0
  -2=Much Worse | 0 | 0

11. Secondary Outcome: Change From Baseline in the Periorbital Aesthetic Appearance Questionnaire (PAAQ) Total Score
Description: The PAAQ consists of 9 questions answered by the participant about their satisfaction with their eye appearance over the past 7 days. Each question is answered using a 5-point scale where: 0=Never (best) to 4=all of the time (worst). The responses to the items on the questionnaire were converted to a 100-point Rasch transformed scale score with 0 (best) to 100 (worst). Lower scores indicate higher satisfaction. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Prior to Treatment) to End of Study (BELKYRA Treatment: Up to Month 11; Non-BELKYRA Treatment: Up to Month 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BELKYRA Treatment | Non-BELKYRA Treatment
Number analyzed (Participants) | 13 | 45
score on a scale
  Baseline | 55.56 (18.215) | 59.69 (17.753)
  Change from Baseline to End of Study | -27.56 (19.394) | -34.07 (24.578)
Statistical Analysis 1: Comparison: BELKYRA Treatment; Test type: Other — The data was analyzed using Paired t-test. If normality was not met, then the Wilcoxon signed-rank test was used; p = 0.0005, Paired t-test/Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: Non-BELKYRA Treatment; Test type: Other — The data was analyzed using Paired t-test. If normality was not met, then the Wilcoxon signed-rank test was used; p < 0.0001, Paired t-test/Wilcoxon Signed Rank Test

ADVERSE EVENTS:
Time Frame: From first dose of study treatment to End of Study (BELKYRA Treatment: Up to Month 11; Non-BELKYRA Treatment: Up to Month 5)
Description: All-cause Mortality: All enrolled participants. Serious Adverse Events and Other Adverse Events: Full Analysis Population included all participants who had met all eligibility criteria at the screening visit and received any product used as treatment in this study.
Arm/Group | BELKYRA Treatment | Non-BELKYRA Treatment
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/45
Other Adverse Events (participants affected / at risk) | 9/13 | 20/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BELKYRA Treatment (N=13) | Non-BELKYRA Treatment (N=45)
Oedema (General disorders) | 4 | 0
Pain (General disorders) | 3 | 0
Injection site reaction (General disorders) | 0 | 2
Nodule (General disorders) | 0 | 2
Cyst (General disorders) | 0 | 1
Injection site bruising (General disorders) | 0 | 1
Injection site pain (General disorders) | 1 | 0
Injection site swelling (General disorders) | 1 | 0
Mass (General disorders) | 0 | 1
Swelling (General disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Herpes simplex (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Post procedural cellulitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 0 | 4
Contusion (Injury, poisoning and procedural complications) | 2 | 1
Injury of conjunctiva (Injury, poisoning and procedural complications) | 0 | 1
Dysaesthesia (Nervous system disorders) | 3 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 2
Brow ptosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Salivary gland pain (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/49/NCT03712449/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT03712449/SAP_001.pdf